CLINICAL TRIAL: NCT02020759
Title: Cerebral Microemboli in Critically Ill Patients Undergoing Venoarterial Extracorporeal Membrane Oxygenation
Brief Title: Cerebral Microemboli in Venoarterial ECMO Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Gabor Erdoes, Dr Gabor Erdoes, Medical University of Vienna
Other Study IDs: 1557/2013
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Complication of Extracorporeal Membrane Oxygenation; Cerebral Microembolism; Cerebral Perfusion
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient on ECMO: Neurological monitoring with transcranial Doppler ultrasound
  Interventions: Device: Transcranial Doppler Ultrasound
- Healthy subjects: Neurological monitoring with transcranial Doppler ultrasound
  Interventions: Device: Transcranial Doppler Ultrasound
- ICU patients: Neurological monitoring with transcranial Doppler ultrasound
  Interventions: Device: Transcranial Doppler Ultrasound

INTERVENTIONS:
Device: Transcranial Doppler Ultrasound — Transcranial Doppler Ultrasound is used to monitor cerebral microembolism

SUMMARY:
Extracorporeal membrane oxygenation (ECMO) is progressively used in critically ill patients with cardiac or respiratory failure as a bridging option for potential organ recovery. However, ECMO survivors often suffer from poor neurocognitive outcome due to neurological complications such as microembolic (ME) strokes.

In venoarterial (va) ECMO circuits the pulmonary circulation, which usually serves as microembolic filter, may be bypassed and generated ME are prone to reach the brain in substantial amounts and potentially impair cerebral integrity. Although patient exposure to cerebral ME has been thoroughly investigated in cardiopulmonary bypass procedures, there is only limited research on cerebral ME in patients undergoing ECMO therapy.

The primary study goal of this study is to determine the load and nature of cerebral ME in critically ill patients under va-ECMO support. We also aim to compare the results to measurements in healthy subjects und intensive care unit (ICU) patients without extracorporeal support to get a better impression on the relevance of ME generation during ECMO support.

DETAILED DESCRIPTION:
The addition of ICU patients was made according to reviewer suggestions after an initial submission to a medical journal.

ELIGIBILITY:
Inclusion Criteria (for patients):

* Intensive care patients with cardiac or respiratory failure under va-ECMO therapy
* Age > 18 yrs.
* Signed informed consent

Exclusion Criteria:

* use of any other extracorporeal device including venovenous (vv) ECMO
* continuous renal replacement therapy
* medical history of severe mitral or aortic stenosis
* medical history of severe mitral or aortic regurgitation
* medical history of carotid stenosis > 70 %
* septicaemia
* medical history of vascular dementia or Alzheimer's disease
* inclusion in an other clinical study
* gravidity
* allergy against materials of one of the medical device used in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of three patient groups with all receiving transcranial Doppler exam: 1. patients undergoing ECMO therapy in the ICU; 2. healthy volunteers, and 3. critically ill controls (patients on the ICU without ECMO)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cerebral embolic load | 30 minutes
  Cerebral embolic load (solid and gaseous) is measured in a 30 minutes-interval during ECMO usage

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Erdoes, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kietaibl C, Horvat Menih I, Engel A, Ullrich R, Klein KU, Erdoes G. Cerebral microemboli during extracorporeal life support: a single-centre cohort study. Eur J Cardiothorac Surg. 2021 Dec 27;61(1):172-179. doi: 10.1093/ejcts/ezab353. PMID 34406372